CLINICAL TRIAL: NCT02684916
Title: Effectiveness of Chiropractic Manipulation Treatment Versus Placebo Manipulation on Children Aged 7-14 Years With Headache and Musculoskeletal Problems. A Randomized Clinical Trial
Brief Title: Chiropractic Treatment for Headache Among Children Aged 7-14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Institute of Chiropractic and Clinical Biomechanics (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1504
Record Dates: First submitted 2016-02-03; First posted 2016-02-18 (Estimated); Last update posted 2020-03-09 (Actual); Status verified 2018-04

CONDITIONS: Chronic Headache
Keywords: Chiropractic spinal manipulation; Children; Pediatric; Headache
MeSH Terms: conditions — Headache Disorders; Headache

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chiropractic treatment (Experimental): Visit with active treatment.
  Interventions: Procedure: Chiropractic treatment
- Placebo (Placebo Comparator): Visit without active treatment.
  Interventions: Procedure: Placebo

INTERVENTIONS:
Procedure: Chiropractic treatment — The child receives chiropractic manipulation treatment in the neck and in the spine and pelvis according to individual needs. They also receive a written list of general advice regarding lifestyle and habits.
  The parents and the child are unaware of group allocation.
  Arms: Chiropractic treatment
Procedure: Placebo — Non-therapeutic placebo treatment: a broad non-specific contact outside the spinal column is taken on subject's scapula and gluteal region lying in a side posture position, on the scapulae in a prone position and on trapezius muscles in a sitting position. In those positions the chiropractor pushes in a non-intentional and non- therapeutic directional line with a low-amplitude, low velocity push maneuver. All contacts are performed without soft tissue pre-tension and gentle contact, to insure that no joint cavitation occurs. To obtain a noise that many people associate with a chiropractic spinal adjustment, a de-activated Activator Instrument is used on the arm of the chiropractor to give a click-sound. General advice on lifestyle and habits is handed out to the placebo group as well.
  Arms: Placebo

SUMMARY:
The primary aim of the study is to assess the effectiveness of chiropractic manipulation treatment versus placebo treatment in children suffering from headache for more than six months.

DETAILED DESCRIPTION:
The study is a two-armed parallel, randomized controlled clinical trial where children suffering from chronic headache and at the same time having one or more biomechanical dysfunctions of the spine are randomized to either chiropractic manipulation treatment or placebo manipulation treatment.

The outcome is based on weekly sms responses collecting the number of days with headache the past week, intensity of headache and use of medication for headache. These are answered four weeks prior to initiation of treatment and 16 weeks thereafter. After the 16 weeks follow-up, a final questionnaire is completed including information about the course and the present headache status.

The primary outcome is the number of days with headache. Secondary outcomes are intensity of headaches and use of medication for headache.

Covariates are collected via baseline questionnaires on patient demographics; medical history; factors known to initiate, worsen or ease the headache; prevalence of headache in the nearest family; and behavioral patterns known to influence headache.

ELIGIBILITY:
Inclusion Criteria:

* Headaches for at least half a year.
* Headache for at least 4 days pr. month.
* At least one musculoskeletal dysfunction as identified by an experienced chiropractor as a movement restriction in one or more of the spinal joints and painful on manual palpation suitable for chiropractic manipulation treatment at the time of the initial screening.
* Able to report information on headache via cell phone either by him- or herself or with help from the parents.

Exclusion Criteria:

* Contraindications for chiropractic treatment
* Ongoing treatment for headache at another practitioner, except medical treatment 3 months prior to inclusion.
* Lack of reporting baseline data via sms 4 weeks prior to inclusion.
* Acute neck or head trauma during the trial period which is estimated to influence the headache

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Difference in number of days per week with headache over four months analyzed as repeated measures with end-point at four months. | Assessed weekly for a period of four months.
  Patient or parent reported via sms-service.

SECONDARY OUTCOMES:
Intensity of headache, graded on a 0-10 scale, where 10 is the worst, over four months analyzed as repeated measures with end-point at four months. | Assessed weekly for a period of four months.
  Patient or parent reported via sms-service.
Use of medicine the past week due to headache over four months analyzed as repeated measures with end-point at four months. | Assessed weekly for a period of four months.
  Patient or parent reported via sms-service.
Improvement on a seven point Likert scale (from 'totally recovered' to 'worse than ever') assessed at four months. | Assessed at the end of four months follow-up.
  Patient or parent reported via sms-service.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne L. Rosing, D.C., MSC, Principal Investigator — Nordic Institute of Chiropractic and Clinical Biomechanics
Locations (1):
- Kiropraktisk Center og Børneklinik, Brønderslev, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lynge S, Vach W, Dissing KB, Hestbaek L. Potential effect modifiers for treatment with chiropractic manipulation versus sham manipulation for recurrent headaches in children aged 7-14 years: development of and results from a secondary analysis of a randomised clinical trial. Chiropr Man Therap. 2023 Jul 11;31(1):20. doi: 10.1186/s12998-023-00492-2. PMID 37434189
- [Derived] Dissing KB, Vach W, Lynge S, Christensen HW, Hestbaek L. Description of recurrent headaches in 7-14-year-old children: Baseline data from a randomized clinical trial on effectiveness of chiropractic spinal manipulation in children with recurrent headaches. Chiropr Man Therap. 2023 Jan 30;31(1):5. doi: 10.1186/s12998-023-00479-z. PMID 36717833
- [Derived] Lynge S, Dissing KB, Vach W, Christensen HW, Hestbaek L. Effectiveness of chiropractic manipulation versus sham manipulation for recurrent headaches in children aged 7-14 years - a randomised clinical trial. Chiropr Man Therap. 2021 Jan 7;29(1):1. doi: 10.1186/s12998-020-00360-3. PMID 33413519
- [Derived] Lynge S, Hartvigsen J, Christensen HW, Vach W, Hestbaek L. Effectiveness of chiropractic manipulation versus sham manipulation on recurrent headaches in children aged 7-14 years, Protocol for a randomized clinical trial. Chiropr Man Therap. 2019 Aug 23;27:40. doi: 10.1186/s12998-019-0262-y. eCollection 2019. PMID 31462990